CLINICAL TRIAL: NCT06847555
Title: Phase I-II Clinical Study of Taurine for External Use in the Prevention and Treatment of Acute Radiation Skin Injury
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Han Xi Zhao, Deputy Chief Physician, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GTEBC-2024
Record Dates: First submitted 2024-08-21; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: To Evaluate the Safety of Taurine in Preventing Acute Radiation Skin Injury Induced by Adjuvant Radiotherapy in Breast Cancer Patients
MeSH Terms: interventions — Radiation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Taurine solution ARM (Experimental): Taurine solution was sprayed to the irradiated area three times a day from 1 day before the start of radiotherapy to 2 weeks after the end of radiotherapy. It is important to spray each time freshly prepared and at a fixed time each morning, noon and evening to ensure continuous contact between the drug and the skin.
  Interventions: Radiation: Radiation

INTERVENTIONS:
Radiation: Radiation — Tumor radiotherapy is a method of treating malignant tumors by using radioactive rays such as alpha, beta, gamma rays produced by radioactive isotopes and x-rays, electron rays, proton beams and other particle beams produced by various x-ray therapy machines or accelerators.

SUMMARY:
Acute radiation skin injury is the most common side effect of radiation therapy in patients with chest tumors, which can be manifested as erythema, dry peeling, wet peeling, and severe ulcers.

Even with current advanced radiotherapy techniques, such as intensity-modulated reverse radiation therapy (IMRT), about one-third of patients develop grade 2 or higher skin damage during radiotherapy. Radiation skin damage can cause discomfort to patients, thus affecting their daily life and reducing their quality of life. In severe cases, it can even reduce the efficacy due to prolonged treatment time. Therefore, prevention and treatment of acute radiation skin injury is a difficult problem to be solved urgently in clinical practice.

Even with current advanced radiotherapy techniques, such as intensity-modulated reverse radiation therapy (IMRT), about one-third of patients develop grade 2 or higher skin damage during radiotherapy. Radiation skin damage can cause discomfort to patients, thus affecting their daily life and reducing their quality of life. In severe cases, it can even reduce the efficacy due to prolonged treatment time. Therefore, prevention and treatment of acute radiation skin injury is a difficult problem to be solved urgently in clinical practice.

From previous studies, we found that taurine is an active substance that regulates normal physiological activities of the body and is widely distributed in various tissues and organs of the body. This substance has many advantages. Many previous studies have shown that taurine also has a wide range of biological functions such as anti-inflammatory, analgesic, maintaining osmotic pressure balance, improving visual function, regulating blood sugar, nerve conduction, endocrine activity, regulating lipid digestion and absorption, increasing cardiac contractility, improving immunity, enhancing cell membrane antioxidant capacity, protecting myocardial cells, etc.

Considering the multiple medical values of taurine and its safety, we intend to conduct a phase I-II clinical study of taurine for external use in the prevention and treatment of acute radiation skin injury for radiation skin injury, with the study period from January 25,2024 to January 25,2027. The purpose is to evaluate the safety of taurine in the prevention and treatment of acute radiation skin injury in breast cancer patients after adjuvant radiotherapy. Possible benefits: Reduce the incidence and severity of radiation skin damage.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients scheduled for conventional fractionated adjuvant
* radiotherapy.
* 18 years or older
* ECOG score 0-1
* No previous history of other neoplasms.
* No previous chest radiotherapy.
* Heart, lung function, liver function and kidney function were within normal range.
* Voluntary informed consent.

Exclusion Criteria:

* Pregnant or lactating women, women in childbearing years who do not use effective contraception；
* Patients with mental disease or nervous system disease, unable to clearly describe treatment response (such as cerebrovascular accident sequela);
* Those who have serious heart, liver, kidney and other organ diseases or diabetes and are not expected to complete the treatment plan;
* serious, uncontrolled diseases and infections;
* Pregnant or lactating patients.
* Allergic to taurine and any of its components.
* Has participated in other clinical trials.
* knot tissue disease
* active hepatitis
* Obvious diseases that the investigator considers should be excluded from this study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-05-25 (Estimated); Primary Completion 2027-09-25 (Estimated); Study Completion 2027-09-25 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate of radiation skin injury | baseline and up to 14 days post-treatment
  Assessed by RTOG Grading criteria for acute radiation skin damage （0-4level）

SECONDARY OUTCOMES:
Change in STAT criteria subjective symptom scores during treatment | baseline and up to 14 days post-treatment
  Subjective symptom scores were recorded weekly with STAT table，contains burning, itching, pulling, pain and other discomfort

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Cancer Hospital, Jinan, Shandong, China